CLINICAL TRIAL: NCT01460745
Title: A Retrospective Review of Liver Resection Rate in Metastatic Colorectal Cancer Patients Following Downsizing Treatment With Chemotherapy Plus Cetuximab in Normal UK National Health Service Clinical Practice
Acronym: RESECT
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Limited, UK (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR062202-546
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Erbitux; CRC; mCRC; Liver; Metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
This study is a multi-centre retrospective observational research study which will be conducted in UK centres with specialised liver surgical services.

The study will involve retrospective review of medical records of patients with metastatic colorectal cancer (mCRC) with metastases confined to the liver, defined locally as unresectable without downsizing therapy at first review by a Hepatobiliary Multi Disciplinary Team (HPB MDT). Erbitux is available for use in combination with chemotherapy as a downsizing treatment for patients with previously unresectable metastases.

The study aims to examine liver resection rates achieved in normal clinical practice in order to inform National Health Service (NHS) clinical and policy decision making and to further understanding of how cetuximab is used in a standard clinical setting. This study intends to estimate the proportion of patients with unresectable liver metastases who undergo liver resection following downsizing treatment with chemotherapy plus cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had mCRC and metastases confined to the liver
* Patients in whom downsizing regimens are recommended
* Patients in whom downsizing treatment included cetuximab
* Patients referred to Hepatobiliary Multi Disciplinary Team (HPB MDT) between 01.01.2010-31.03.2011

Exclusion Criteria:

* Patients who are considered to have immediately resectable liver metastases as determined by the HPB MDT
* Patients who are considered to have never resectable liver metastases as determined by the HPB MDT
* Patients who were aged less than 18 at date of initiation of cetuximab
* Patients who are enrolled in a clinical trial during the data collection period
* Patients who are receiving private healthcare for the treatment of mCRC
* According to Summary of Product Characteristics (SmPC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who undergo liver resection following downsizing chemotherapy with or without Erbitux | 7 months

SECONDARY OUTCOMES:
Percentage of liver resection outcomes R0, R1 and R2 | 7 months
  The liver resection outcomes are defined as follows: R0: Absence of microscopic tumor invasion of the resection margins (tumour free margin ≥ 1mm); R1: Presence of microscopic tumor invasion of the resection margins (tumour free margin 0mm); R2: Presence of macroscopic positive margin after resection

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serpno Limited, UK, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (5):
- United Kingdom (5):
  - Merck Serono Research Site, Bristol
  - Merck Serono Research Site, Liverpool
  - Merck Serono Research Site, London
  - Merck Serono Research Site, Manchester
  - Merck Serono Research Site, Southampton

REFERENCES:
- [Result] Malik H, Khan AZ, Berry DP, Cameron IC, Pope I, Sherlock D, Helmy S, Byrne B, Thompson M, Pulfer A, Davidson B. Liver resection rate following downsizing chemotherapy with cetuximab in metastatic colorectal cancer: UK retrospective observational study. Eur J Surg Oncol. 2015 Apr;41(4):499-505. doi: 10.1016/j.ejso.2015.01.032. Epub 2015 Feb 7. PMID 25703078